CLINICAL TRIAL: NCT05913908
Title: Early Feasibility Study of the DUO Transcatheter Tricuspid Coaptation Valve System in Patients With Tricuspid Regurgitation
Brief Title: EFS of the DUO System for Tricuspid Regurgitation
Acronym: TANDEM II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CroiValve Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV006
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Tricuspid Regurgitation; Tricuspid Valve Insufficiency; Tricuspid Valve Disease; Heart Valve Diseases
Keywords: Transcatheter; Coaptation Valve; TR; SVC; Tricuspid
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the DUO Transcatheter Tricuspid Coaptation Valve System (DUO System)
  Interventions: Device: DUO Transcatheter Tricuspid Coaptation Valve System

INTERVENTIONS:
Device: DUO Transcatheter Tricuspid Coaptation Valve System — Reduction of tricuspid regurgitation through a transcatheter approach
  Other Names: DUO System

SUMMARY:
The study is an early feasibility study to measure individual patient clinical outcomes and effectiveness, evaluate the safety and function of the DUO Transcatheter Tricuspid Coaptation Valve System (DUO System).

DETAILED DESCRIPTION:
Multi-center, prospective, non-randomized, investigational, and pre-market. Data collected in this clinical study will include safety and function of the investigational system as well as up to 5 year clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of severe or greater tricuspid regurgitation as determined by the Echo Core Lab.
2. Patient is symptomatic despite medical therapy.
3. The local Site Heart Team determines the Patient is appropriate for transcatheter valve intervention.
4. The Patient's anatomy is suitable in the judgment of the Patient Selection Committee.
5. Age ≥18 years
6. The Patient has been informed of the nature of the study and agrees to its provisions and has provided written Informed Consent.

Exclusion Criteria:

1. Patient is currently participating in another clinical investigation that could affect the outcome of this trial.
2. Any previous tricuspid valve intervention that would interfere with the placement of the investigational device.
3. Moderate or greater tricuspid valve stenosis.
4. Severe aortic, mitral and/or pulmonic valve stenosis and/or regurgitation
5. Pacemaker or implantable cardioverter-defibrillator (ICD) leads that would prevent appropriate placement of the investigational device.
6. Need for concomitant surgical or interventional procedure, known at the time of screening (e.g., CABG, Atrial Septal Defect (ASD) repair).
7. Ejection Fraction (EF) <25%
8. Echocardiographic evidence of unstable intracardiac mass, thrombus or vegetation
9. Patient has Systolic Pulmonary Pressure (sPAP) >60 mm Hg
10. Severe hemodynamic instability: cardiogenic shock or the need for inotropic support or Intra-Aortic Balloon Pump (IABP) or other percutaneous ventricular assist devices
11. Severe respiratory instability with continuous use of home oxygen
12. Severe right ventricular dysfunction
13. Untreated clinically significant coronary or carotid artery disease requiring revascularization surgical or interventional PCI.
14. Stroke or transient ischemic event within 90 days prior to the index procedure
15. Acute myocardial infarction within 30 days before the index procedure
16. Renal insufficiency (eGFR <25 ml/min) or currently on chronic dialysis
17. Active endocarditis within 6 months of the index procedure
18. Pulmonary embolism or deep vein thrombosis within the last 6 months
19. Any surgical, interventional, or transcatheter procedure within 30 days prior to the index procedure
20. Hypertrophic cardiomyopathy, restrictive cardiomyopathy or constrictive pericarditis
21. Life expectancy <1 year
22. Active infections requiring current antibiotic therapy
23. Known severe liver disease
24. Is on the waiting list for a transplant or has had a prior heart or lung transplant
25. Known active peptic ulcer or active GI bleed
26. Unable to take anticoagulant therapy
27. Any known major coagulation abnormalities, thrombocytopenia, platelets < 50,000/ml or severe anemia Hb <8 g/dl
28. Known patient is actively abusing drugs
29. Any known sensitivities or allergies to contrast (that cannot be adequately premedicated) and/or the device materials, including nickel and titanium
30. Patients who are pregnant or intend to become pregnant
31. Any condition making it unlikely the Patient will be able to complete all protocol procedures (including compliance with optimal medical therapy and immobility that would prevent completion of 6MWT), follow-up visits, or impact the scientific soundness of the clinical investigation result

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from device or procedure related MAEs | At 30 days
  * Death
  * Reintervention
  * Disabling stroke
  * Myocardial infarction
  * Major access site and vascular complications
  * Severe bleeding
  * Renal failure requiring dialysis
  * Major cardiac structural complications
  * Pulmonary embolism

CONTACTS AND LOCATIONS:
Locations (16):
- United States (13):
  - Dignity Health St. Joseph's Hospital & Medical Center, Phoenix, Arizona
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Ascension Via Christi Research, Wichita, Kansas
  - Allina Health Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University Medical Center/NYPH, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - OhioHealth Research Institute, Columbus, Ohio
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - San Antonio Methodist, San Antonio, Texas
  - Intermountain Health, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Poland (3):
  - Uniwersytetem Medycznym im. Karola Marcinkowskiego w Poznaniu, Poznan, Poznan
  - Narodowym Instytutem Kardiologii Stefana Kardynała Wyszyńskiego - Państwowym Instytutem Badawczym, Warsaw, Warsaw
  - Medical University of Silesia, Katowice